CLINICAL TRIAL: NCT05817643
Title: A Randomized, Open-label, 2-period, Crossover, Pilot Food Effect Study of BMS-984923 in Healthy Older Adult Volunteers
Brief Title: Food Effect Study of BMS-984923 in Healthy Older Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Allyx Therapeutics (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALX-923-103
Record Dates: First submitted 2023-03-24; First posted 2023-04-18 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Under Fed Condition (Active Comparator): Investigational Drug is administered with a meal
  Interventions: Drug: BMS-984923
- Dose Under Fasted Condition (Active Comparator): Investigational Drug is administered after fasting
  Interventions: Drug: BMS-984923

INTERVENTIONS:
Drug: BMS-984923 — Oral capsule

SUMMARY:
This project is developing a novel disease-modifying compound for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate for an effect of food consumption on the pharmacokinetics profile of BMS984923. Safety and tolerability is also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 50 and 80 years, inclusive
* No history of cognitive impairment
* Capable of providing written informed consent and willing to comply with all study requirements and procedures
* Participant is not pregnant, lactating, or of childbearing potential

Exclusion Criteria:

* Body mass index (BMI) >38 kg/m2 or body weight <50 kg.
* Significant cerebrovascular disease
* Any significant neurologic disease
* A current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM V) diagnosis of active major depression, schizophrenia or bipolar disorder
* Clinically significant or unstable medical condition
* Any disorder or medication that could interfere with the absorption, distribution, metabolism or excretion of drugs
* History of cholecystectomy
* History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for hepatitis B surface antigen [HbsAg] or anti-hepatitis C virus [HCV] antibody).
* Use of psychoactive medications
* Use of medications with potential drug-drug interactions
* Use of another investigational agent
* Clinically significant abnormalities in screening laboratories
* Any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale
* Acceptable Geriatric Depression Scale (GDS) score

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 10 days after last dose
  Maximum plasma concentration as determined by pharmacokinetic modeling
Time of Cmax (Tmax) | Up to 10 days after last dose
  Time of Cmax as determined by pharmacokinetic modeling
Area Under the Curve from 0 to 24h (AUC 24h) | Up to 10 days after last dose
  Plasma drug exposure as determined by pharmacokinetic modeling

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAE) | 14 days
  Safety
Safety Laboratory abnormalities | 14 days
  Safety
Electrocardiogram - QT Interval | 14 days
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Post, MD, Principal Investigator — Principal Investigator
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No